CLINICAL TRIAL: NCT05499351
Title: A Single Center, Randomized ,Controlled and Open Clinical Trial to Evaluate the Immunogenicity and Safety of the Booster Immunization With the Third Dose of COVID-19 Vaccine,Inactivated Co -Administration With Influenza Vaccine and Pneumococcal Polysaccharide Vaccine
Brief Title: A Study of Booster Immunization With COVID-19 Vaccine,Inactivated Co -Administration With Influenza Vaccine and Pneumococcal Polysaccharide Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-nCOV-MA4005-BJ
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult group in immunogenicity and safety study of combined immunization (Experimental): 300 participants will be randomly divided into 3 subgroups of 100 people per group, each subject will receive 1 dose of COVID-19 vaccine, 1 dose of influenza vaccine and 1 dose of pneumonia vaccine
  Interventions: Biological: Adult group in immunogenicity and safety study of combined immunization
- Elderly group in immunogenicity and safety study of combined immunization (Experimental): 300 participants will be randomly divided into 3 subgroups of 100 people per group, each subject will receive 1 dose of COVID-19 vaccine, 1 dose of influenza vaccine and 1 dose of pneumonia vaccine
  Interventions: Biological: Elderly group in immunogenicity and safety study of combined immunization
- Adult group in safety observation study of combined immunization (Experimental): 1200 participants will be randomly divided into 2 subgroups of 600 people per group, each subject will receive 1 dose of COVID-19 vaccine, 1 dose of influenza vaccine and 1 dose of pneumonia vaccine
  Interventions: Biological: Adult group in safety observation study of combined immunization
- Elderly group in safety observation study of combined immunization (Experimental): 1200 participants will be randomly divided into 2 subgroups of 600 people per group, each subject will receive 1 dose of COVID-19 vaccine, 1 dose of influenza vaccine and 1 dose of pneumonia vaccine
  Interventions: Biological: Elderly group in safety observation study of combined immunization

INTERVENTIONS:
Biological: Adult group in immunogenicity and safety study of combined immunization — The COVID-19 vaccine was manufactured by Sinovac Research & Development Co., Ltd,and the quadrivalent influenza vaccine and the 23-valent pneumococcal polysaccharide vaccine(PPV23) were manufactured by Sinovac Biotech Co.The COVID-19 vaccine:600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection;The quadrivalent influenza vaccine:15ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection;PPV23:capsular polysaccharides of 23 serotypes of pneumococcus in 0.5 mL of Sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.
  Arms: Adult group in immunogenicity and safety study of combined immunization
Biological: Elderly group in immunogenicity and safety study of combined immunization — The COVID-19 vaccine was manufactured by Sinovac Research & Development Co., Ltd,and the quadrivalent influenza vaccine and the 23-valent pneumococcal polysaccharide vaccine(PPV23) were manufactured by Sinovac Biotech Co.The COVID-19 vaccine:600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection;The quadrivalent influenza vaccine:15ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection;PPV23:capsular polysaccharides of 23 serotypes of pneumococcus in 0.5 mL of Sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.
  Arms: Elderly group in immunogenicity and safety study of combined immunization
Biological: Adult group in safety observation study of combined immunization — The COVID-19 vaccine was manufactured by Sinovac Research & Development Co., Ltd,and the quadrivalent influenza vaccine and the 23-valent pneumococcal polysaccharide vaccine(PPV23) were manufactured by Sinovac Biotech Co.The COVID-19 vaccine:600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection;The quadrivalent influenza vaccine:15ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection;PPV23:capsular polysaccharides of 23 serotypes of pneumococcus in 0.5 mL of Sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.
  Arms: Adult group in safety observation study of combined immunization
Biological: Elderly group in safety observation study of combined immunization — The COVID-19 vaccine was manufactured by Sinovac Research & Development Co., Ltd,and the quadrivalent influenza vaccine and the 23-valent pneumococcal polysaccharide vaccine(PPV23) were manufactured by Sinovac Biotech Co.The COVID-19 vaccine:600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection;The quadrivalent influenza vaccine:15ug hemagglutinin (HA) of each of the four influenza strains in 0.5 mL of sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection;PPV23:capsular polysaccharides of 23 serotypes of pneumococcus in 0.5 mL of Sodium chloride, disodium hydrogen phosphate, sodium dihydrogen phosphate per injection.
  Arms: Elderly group in safety observation study of combined immunization

SUMMARY:
This study is a single center , randomized ,controlled and open-label phase Ⅳclinical trial of the booster immunization with the third dose of inactivated COVID-19 vaccine(CoronaVac)manufactured by Sinovac Research & Development Co.,Ltd. The purpose of this study is to evaluate the immunogenicity and safety of the third dose of COVID-19 vaccine,inactivated (Vero Cell) co-administration with influenza vaccine and pneumococcal polysaccharide vaccine in healthy population aged 18 years and older.

DETAILED DESCRIPTION:
This study is a single center , randomized ,controlled and open-label phase Ⅳclinical trial in healthy adult aged 18 years and older. The purpose of this study is to evaluate the immunogenicity and safety of the third dose of COVID-19 vaccine,inactivated (Vero Cell) co-administration with influenza vaccine and pneumococcal polysaccharide vaccine.The COVID-19 vaccine was manufactured by Sinovac Research &Development Co., Ltd,and the quadrivalent influenza vaccine and 23-valent pneumococcal polysaccharide vaccine(PPV23) were manufactured by Sinovac Biotech Co.A total of 3000 subjects will be enrolled, with 300 aged 18~59years(adult group) and 300 aged 60 years and above(adult group) in the section of immunogenicity and safety of combined immunization ,with 1200 aged 18~59 years(adult group) and 1200 aged 60 years and above(elderly Group) in the section of safety observation study of combined immunization.Each age group will be randomly divided into 3 subgroups of 100 people per group, each subject will receive 1 dose of COVID-19 vaccine, 1 dose of influenza vaccine and 1 dose of pneumonia vaccine in the section of immunogenicity and safety of combined immunization and each age group will be randomly divided into 2 subgroups of 600 people per group, each subject will receive 1 dose of COVID-19 vaccine, 1 dose of influenza vaccine and 1 dose of pneumonia vaccine in the section of safety observation study of combined immunization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 years and above;
* Have been received two doses of inactivated SARS-CoV-2 vaccine(CoronaVac)manufactured by Sinovac Research & Development Co., Ltd at an interval of 6 months or more;
* Participants should be capable of understanding the informed consent form, and such form should be signed prior to enrolment ;
* Proven legal identity;

Exclusion Criteria:

* History of SARS-CoV-2 infection;
* Have been received two doses of inactivated SARS-CoV-2 vaccine(CoronaVac)manufactured by Sinovac Research & Development Co., Ltd at an interval of less than 6 months;
* Have received received any circulating seasonal influenza vaccine;
* Have received any pneumococcal vaccine within 5 years;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* History of uncontrolled epilepsy and other serious neurological diseases such as transverse myelitis, Guillain-Barre syndrome, demyelinating diseases;
* History of fever at the time of vaccination, or acute onset of chronic disease, or severe uncontrolled chronic disease, or acute disease;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Immunogenicity index of seroconversion rate of the neutralizing antibody | 28 days after the booster immunization with the third dose of COVID-19 vaccine
  Seroconversion rate of the neutralizing antibody to live SARS-CoV-2 28 days after the booster immunization with the third single dose of COVID-19 vaccine

SECONDARY OUTCOMES:
Immunogenicity index of seropositivity rate of the neutralizing antibody | 28 days after combined immunization
  Seropositivity rate of the neutralizing antibody to live SARS-CoV-2 28 days after combined immunization
Immunogenicity index of GMT of the neutralizing antibody | 28 days after combined immunization
  GMT of the neutralizing antibody to live SARS-CoV-2 28 days after combined immunization
Immunogenicity index of GMI of the neutralizing antibody | 28 days after combined immunization
  GMI of the neutralizing antibody to live SARS-CoV-2 28 days after combined immunization.
Immunogenicity index of seroconversion rate of 23 pneumonia antibodies | 28 days after single and combined vaccination of 23 valent pneumonia vaccine
  Seroconversion rate of 23 pneumonia antibodies 28 days after single and combined vaccination of 23 valent pneumonia vaccine.
Immunogenicity index of GMC increase of 23 pneumonia antibodies | 28 days after single and combined vaccination of 23 valent pneumonia vaccine
  GMC increase of 23 pneumonia antibodies 28 days after single and combined vaccination of 23 valent pneumonia vaccine
Immunogenicity index of seroconversion rate of 4 influenza antibodies | 28 days after single and combined vaccination
  Seroconversion rate of 4 influenza antibodies 28 days after single and combined vaccination
Immunogenicity index of GMT of 4 influenza antibodies | 28 days after single and combined vaccination
  GMT of 4 influenza antibodies 28 days after single and combined vaccination
Immunogenicity index of GMI of 4 influenza antibodies | 28 days after single and combined vaccination
  GMI of 4 influenza antibodies 28 days after single and combined vaccination
Immunogenicity index of protection rate of 4 influenza antibodies | 28 days after single and combined vaccination
  Protection rate of 4 influenza antibodies 28 days after single and combined vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, Master, Principal Investigator — Beijing Center for Disease Control and Prevention
Locations (1):
- Beijing Centers for Diseases Control and Prevention, Beijing, China